CLINICAL TRIAL: NCT03316768
Title: Measurement of Grip and Pinch Forces Needed for Activities of Daily Living, Work and Prehistoric Stone Tool Production
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 01D23E57.603E53E0
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2018-04

CONDITIONS: Basilar Thumb Arthritis; Wrist Fracture; Measure Pressure Distribution and Resultant Forces Needed
Keywords: grip; pinch; forces; pressure; Tekscan; sensor; ADL; activities of daily living; work requirements; hand biomechanics; forceful precision grip; power grip; hominid; hominin; prehistoric
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Very little is known about the pinch and grip forces that are critical for activities of daily living (ADL) or work. Human success in evolution is a result of the combination of great brain power and great hand ability to accomplish with our hands what our minds can conceive. Prehensile grasp in hominins allowed tool production and today allows us to hold fine instruments to perform surgery or do heavy construction. The strength of our hands is matched against the requirements of the activities we need to perform. The hypothesis of this study is that many tasks have an inherent strength requirement that is independent of the person performing the task. Until recently, direct measurement of the forces has not been possible. Ultra thin sensors along with the software to interpret the information is now available to make this force determination possible. We have 3 primary objectives. The primary objective is to measure pressure distribution and resultant forces needed for 3 categories of ADL and 2 categories of work in normal subjects. The second objective is to perform a similar evaluation of patients with basilar thumb arthritis and after wrist fracture. The third objective is to measure pressure distribution and forces needed for tool production and use.

DETAILED DESCRIPTION:
The study will measure pressures and forces for ADL and simulated work using healthy volunteers. Sixteen volunteers will be chosen over a range of ages but specifically include similar numbers of early adulthood (18-44), middle age (45-65), and elderly (>65). Sixteen volunteers from each age group divided evenly by gender will be selected. Therefore, a total of 48 subjects will be tested, with an even number of male and female performing each of the activities listed above.

Inclusion Critera Volunteers will be recruited through website, personnel, and community contacts. They will be recruited based on age and gender.

Exclusion Criteria Patients will be excluded if they have a history of an inflammatory condition such as rheumatoid arthritis or lupus. They will be excluded if they have symptomatic osteoarthritis of their hands. Additional exclusion criteria will include known neurologic conditions, or prior injury that may be contributing to weakness or atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* At least 18 years old
* Willing to participate in the study

Exclusion Criteria:

* History of an inflammatory condition such as rheumatoid arthritis or lupus
* Symptomatic osteoarthritis of their hands
* Known neurologic condition
* Prior injury that may be contributing to weakness or atrophy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited through website, personnel, and community contacts. They will be recruited based on age and sex. Helsinki approval will be obtained before recruiting patients. Informed consent will be obtained.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | one day
  Grip Strength